CLINICAL TRIAL: NCT05361174
Title: A Phase 1/2, Open-label Study of PD-1 Knockout Tumor-infiltrating Lymphocytes (IOV-4001) in Participants With Unresectable or Metastatic Melanoma or Stage III or IV Non-small-cell Lung Cancer
Brief Title: A Study to Investigate the Efficacy and Safety of an Infusion of IOV-4001 in Adult Participants With Unresectable or Metastatic Melanoma or Stage III or IV Non-small-cell Lung Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Iovance Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IOV-GM1-201
Record Dates: First submitted 2022-04-29; First posted 2022-05-04 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Unresectable Melanoma; Metastatic Melanoma; Stage III Non-small Cell Lung Cancer; Stage IV Non-small Cell Lung Cancer
Keywords: Tumor Infiltrating Lymphocytes; TIL; Unresectable Melanoma; Metastatic Melanoma; Stage III Non-small-cell lung cancer; Stage IV Non-small-cell lung cancer; PD-1 Knockout; Cell Therapy; Autologous Adoptive Cell Therapy; Cellular Immuno-therapy; IL-2; Non Small Cell Lung Cancer; NSCLC; Second line Lung Cancer; Bronchial Neoplasms; Carcinoma; Lung Disease; Metastatic Lung Cancer; Metastatic Non Small Cell Lung Cancer; Lung Carcinoma; PD-L1; Stage IV Cancer; Stage IV Lung Cancer; Stage IV NSCLC; Systemic Therapy; 2nd line therapy; Second line therapy; CPI; Check point inhibitor; Metastatic NSCLC; NSCLC Recurrent; Recurrent Lung Cancer; Recurrent Lung Carcinoma; Autologous Adoptive Cell Transfer; Melanoma; Lifileucel; Stage III Melanoma; Stage IV Melanoma; Skin cancer; Skin cancer types; Malignant melanoma
MeSH Terms: conditions — Melanoma; Carcinoma, Non-Small-Cell Lung; Bronchial Neoplasms; Carcinoma; Lung Diseases; Lung Neoplasms; Neoplasms; Skin Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): Participants with unresectable or metastatic melanoma
  Interventions: Biological: IOV-4001
- Cohort 2 (Experimental): Participants with Stage III or IV non-small-cell lung cancer
  Interventions: Biological: IOV-4001

INTERVENTIONS:
Biological: IOV-4001 — A tumor sample is resected from each participant and cultured ex-vivo to manufacture IOV-4001. After lymphodepleting chemotherapy including cyclophosphamide and fludarabine, participant is infused with IOV-4001, and followed by IL-2.

SUMMARY:
This is a study to investigate the efficacy and safety of an infusion of IOV-4001 in adult participants with unresectable or metastatic melanoma or advanced non-small-cell lung cancer (NSCLC).

DETAILED DESCRIPTION:
This study is the first-in-human study of IOV-4001, a genetically modified autologous tumor- infiltrating lymphocytes (TIL) product. IOV-4001 is expected to have antitumor activity through its capacity to directly target and kill tumor cells in a manner that is similar to non-genome-edited TIL, but with the potential for enhanced antitumor activity due to disruption of PDCD1, the gene for programmed cell death protein-1 (PD-1).

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have a confirmed diagnosis of Stage IIIC, IIID, or IV unresectable or metastatic melanoma or Stage III or IV NSCLC.
2. Participants who have received the following previous therapy:

   1. Cohort 1 (Melanoma): Participants who have progressed within 12 weeks of last dose of anti-PD-1/PD-L1 blocking antibody and received BRAF/MEK inhibitor in those with BRAF mutations.
   2. Cohort 2 (NSCLC): Participants who should have received no more than 3 prior lines of therapy and:

      * those without oncogene-driven tumors: Have progressed within 12 weeks after last dose of anti-PD-1/PD-L1 blocking antibody
      * those with oncogene-driven tumors: Have progressed during/after ≥1 targeted therapy AND either:

        * platinum doublet chemotherapy
        * Or within 12 weeks after last dose of anti-PD-1/PD-L1 blocking antibody
3. Participants who have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
4. Participants who is assessed as having at least one resectable lesion.
5. Participants who have at least one measurable lesion, following resection of the lesion for IOV-4001 generation.
6. Participants who have adequate organ function.
7. Cardiac function test required.
8. Pulmonary function test may be required.
9. Participants of childbearing potential or those with partners of childbearing potential must be willing to practice an approved method of highly effective birth control during treatment and up to 12 months.
10. Participants who are >70 years of age may be allowed to enroll after the investigator discusses with the medical monitor.

Exclusion Criteria:

1. Participants who have melanoma of uveal/ocular origin.
2. Participants who have symptomatic untreated brain metastases.
3. Participants who have had a history of allogeneic organ transplant or any form of cell therapy involving prior conditioning chemotherapy within the past 20 years.
4. Participants who require systemic steroid therapy 10 mg/day prednisone or another steroid equivalent dose.
5. Participants who have any form of primary immunodeficiency.
6. Participants who have another primary malignancy within the previous 3 years.
7. Participants who have received or will receive a live or attenuated vaccination within 28 days prior to the start of the NMA-LD.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2022-07-20 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Phase I: Safety of IOV-4001 | Up to 1 Year or depending on when the recommended phase 2 dose is determined
  The safety of IOV-4001 will be assessed based on the totality of dose-limiting toxicity (DLT) and adverse event (AE) data collected during this phase
Phase 2: Objective Response Rate (ORR) | Up to 60 months
  To evaluate the proportion of participants who have a confirmed complete response (CR) or partial response (PR) per RECIST v1.1 as assessed by the investigator

SECONDARY OUTCOMES:
CR Rate | Up to 60 months
  To evaluate the proportion of participants who have a confirmed CR per RECIST v1.1 as assessed by the investigator
Duration of Response (DOR) | Up to 60 months
  To evaluate the duration from the time that criteria are met for CR or PR per RECIST v1.1 as assessed by the investigator until disease progression or death due to any cause
Disease Control Rate (DCR) | Up to 60 months
  To evaluate the percentage of participants with a best overall confirmed response of CR or PR at any time plus stable disease (SD) per RECIST v1.1 as assessed by the investigator
Progression-free Survival (PFS) | Up to 60 months
  To evaluate the time from the date of IOV-4001 infusion until disease progression per RECIST v1.1 as assessed by the investigator or death due to any cause
Overall Survival (OS) | Up to 60 months
  To evaluate the time from the date of IOV-4001 infusion to death due to any cause.
Safety and Tolerability of IOV-4001 | Up to 60 months
  This will be characterized by the severity, seriousness, relationship to study treatment, and characteristics of treatment-emergent adverse events (TEAEs).
Feasibility of IOV-4001 | Up to 60 months
  This will be assessed by the proportion of participants who had tumor harvested and were treated without manufacturing delay or failure.

CONTACTS AND LOCATIONS:
Overall Officials: Iovance Biotherapeutics Study Team, Study Director — Iovance Biotherapeutics
Locations (10):
- United States (10):
  - The Angeles Clinic and Research Institute, Los Angeles, California
  - Sylvester Comprehensive Cancer Center, Miami, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - The University of Kansas Cancer Center, Westwood, Kansas
  - University of Louisville, Louisville, Kentucky
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Cincinnati, Cincinnati, Ohio
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Medical College of Wisconsin, Milwaukee, Wisconsin